CLINICAL TRIAL: NCT01288963
Title: The High-Dose Aldesleukin (IL-2) "SELECT" Trial: A Prospective Tissue Collection Protocol to Investigate Predictive Models of Response to High-Dose IL-2 Treatments in Patients With Advance Melanoma
Brief Title: IL-2 "SELECT" Tissue Collection Protocol in Patients With Advanced Melanoma
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David McDermott, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 09-333
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Malignant Melanoma
Keywords: melanoma; IL-2; Aldesleukin
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IL-2 subjects: Subjects receiving IL-2 for advanced melanoma
  Interventions: Drug: IL-2

INTERVENTIONS:
Drug: IL-2 — Observation only
  Other Names: aldesleukin

SUMMARY:
The purpose of this study is to determine which participants with melanoma have a better response to IL-2 and to identify markers that may predict response to IL-2 by collecting participant information (for example; cancer diagnosis and history, prior treatments for cancer, etc.) blood and tumor samples prior to treatment and tumor measurements after treatment.

DETAILED DESCRIPTION:
Original tumor slides will be collected to identify tumor markers that may predict responses to treatment. Blood samples will be obtained prior to treatment with IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma that is metastatic or unresectable
* Eligible to receive high-dose IL-2
* Tissue block available with adequate tumor to perform RNA extraction and DASL analysis

Exclusion Criteria:

* Prior immunotherapy for unresectable or metastatic disease
* Untreated brain metastases, leptomeningeal disease, or seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled on DF/HCC Protocol 06-149
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
To determine if DASL subclassification can identify a group of patients with advanced melanoma who are significantly more likely to respond to high dose IL-2 based on therapy than the historical 16% response rate in an unselected patient population | 2 years

SECONDARY OUTCOMES:
To validate the usefulness of serum fibronectin and VEGF levels as negative predictors of response | 2 years
To explore the predictive value of several genetic polymorphisms associated with immune function | 2 years
To explore the predictive value of BRAF^V600E mutational status as a predictor of response and benefit to high dose IL-2 | 2 years
To explore the relationship of serum fibronectin and VEGF levels with the molecular signature of immune responsiveness in patients with advanced melanoma receiving high-dose IL-2 in order to identify specific cohorts with dramatic differences in response | 2 years
To identify new proteins or patterns of gene expression that might be associated with high-dose IL-2 responsiveness in order to further narrow the application of IL-2 therapy to those who will benefit the most | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States